CLINICAL TRIAL: NCT04866264
Title: Electronic-Nutrition-Optimizer for Personalized Prevention
Acronym: eNO
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Heike Bischoff-Ferrari (Other)
Responsible Party: Sponsor-Investigator, Heike Bischoff-Ferrari, Director, Geriatric Clinic, University Hospital Zurich, University of Zurich
Organization: University of Zurich (Other)
Allocation: Non-Randomized | Model: Crossover | Masking: None | Purpose: Other
Other Study IDs: 2019-02379
Record Dates: First submitted 2021-04-01; First posted 2021-04-29 (Actual); Last update posted 2024-08-07 (Actual); Status verified 2024-08

CONDITIONS: Diabetes; Hypertension; Frailty; Dementia; Cardiovascular Diseases
Keywords: Mediterranean Diet; MIND Diet; Healthy Aging
MeSH Terms: conditions — Diabetes Mellitus; Hypertension; Frailty; Dementia; Cardiovascular Diseases

STUDY DESIGN:
Intervention Model Description: Pilot study (exploratory case-crossover study) for user feasibility and validation of the eNutrition Optimizer
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Outpatient Group (Active Comparator): After signing the informed consent, outpatients will be invited for a clinical baseline visit at the Center on Aging and Mobility (CAM), where they will complete the dietary assessment with the eNutrition optimizer at the CAM guided by the study physicians, who will also interpret the immediate results and recommendations produced by the tool to the study participant.
  For validating the eNutrition-Optimizer tool, participants will be asked to report their dietary intake in the past 24h during a "24-h diet recall phone call" conducted by a trained interviewer on random days (weekday and weekend), so the participant cannot prepare or alter their habits. This 24h diet recall phone calls will be performed 4 times during the second half of the follow-up (month 4 to 6). In addition participants will complete the System Usability Scale at baseline and the subjective effectiveness questionnaire at month 6.
  Interventions: Device: eNutrition Optimizer
- Inpatient Group (Active Comparator): After signing the informed consent, inpatients (Senior trauma center/heart surgery) will do the dietary assessment with the eNutrition optimizer with supervision of a trained study physician to assess user feasibility in the inpatient setting. In addition they will have a follow-up phone call at month 3 to 6 to assess the subjective effectiveness of the eNO.
  Interventions: Device: eNutrition Optimizer

INTERVENTIONS:
Device: eNutrition Optimizer — The eNutrition optimizer is based on the electronic food frequency questionnaire (FFQ) used in the multicentre randomized controlled trail DO-HEALTH [56] developed by the CAM. The FFQ is split up in sections of 33 food groups and contains 216 items. It asks the user on the relative frequency of consumption of the different foods showing a picture of the food in the portion size of interest. Within the eNutrition Optimizer, the FFQ will be extended to create an output of the user's adherence to the Mediterranean diet, the MIND diet and the adherence with the current dietary recommendations for micro- and macronutrients provided by the Swiss Society for Nutrition and the DACH-references, compare it to the DO-HEALTH population and give recommendations on how to improve the score.

SUMMARY:
This study aims to develop and validate a tool for immediate nutrition assessment and to test its user feasibility in routine clinical practice for health promotion.

DETAILED DESCRIPTION:
Small changes in diet have been shown to have an important impact on health and the risk of age-related chronic diseases, such as cardiovascular disease, diabetes, frailty and dementia. However, this knowledge has not yet been implemented into routine clinical practice, because practical tools that allow a comprehensive nutrition assessment in the clinical care setting are missing. In addition, doctors are generally not educated in giving nutritional advice to patients. In this pilot project, we aim to push forward and enable the potential of nutrition as a core primary prevention strategy for people at risk of developing chronic diseases. This will be achieved by using, as a stepping stone, the electronic 216-food-item food frequency questionnaire which was developed for the European DO-HEALTH study and was tested in over 2000 adults. The investigators want to extend this tool to not only capture the personal dietary intake, but also to produce an immediate report, comparing the personal diet to the Mediterranean and MIND diet patterns and providing a patient's intake of protein and other nutrients. The report will additionally indicate the patient's diet-related, personalized risks of cardio-vascular disease, diabetes, frailty and cognitive decline, and recommend dietary changes to reduce these risks.

ELIGIBILITY:
Inclusion Criteria:

1. Stable inpatients from the Department of heart surgery, or Center for senior trauma patient at the university hospital Zurich (inpatient group)
2. Ambulatory volunteers who can visit the center for aging and mobility (CAM) independently ("outpatients" group)
3. ≥50 years

Exclusion Criteria:

1. If already involved in another ongoing interventional clinical trial, except an interaction with this intervention can be excluded
2. People with an impaired short-term memory (MMSE <24)
3. Patients following a specific diet recommended by a medical professional, due to diseases such as diabetes, chronic diseases of the gastrointestinal tract, severe kidney disease, or patients allergic to the main components of the Mediterranean diet/MINDdiet (olive oil, nuts)
4. Outpatients: HbA1C ≥6.5% Inpatients: HbA1C ≥6.5% or diagnosed diabetes mellitus if HbA1C is not available in KISIM
5. BMI > 30 kg/m2
6. Individuals per se not willing to change diet
7. Instable clinical conditions (e.g. acute infection) at enrolment
8. Patients with active cancer (except non-melanoma skin cancer) or current cancer treatment or any other advanced severe disease
9. Living in a nursing home and/or receiving prepared meals (i.e. usually not eating home cooked meals)
10. Inability to read and or speak German necessary to understand the instructions

Min Age: 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 88 (Actual)
Dates: Start 2021-11-11 (Actual); Primary Completion 2024-05-23 (Actual); Study Completion 2024-05-23 (Actual)

PRIMARY OUTCOMES:
Perception questionnaire using system usability scale | Baseline
  Feasibility Study (in- and outpatient group) Scale from 1 to 5, indicating 1 "not true", 5 "very true"
Subjective effectiveness questionnaire of eNutrition Optimizer | month 3 to 6
  Feasibility Study (in- and outpatient group) Scale from 1 to 5, indicating 1 "not true", 5 "very true"

SECONDARY OUTCOMES:
24h diet recalls | month 4 to 6
  Validation Study (outpatient group)
blood marker Non-HDL cholesterol (mmol/l) | 6 months
  Validation Study (outpatient group)
blood marker HDL cholesterol (mmol/l) | 6 months
  Validation Study (outpatient group)
blood marker Triglycerides (mmol/l) | 6 months
  Validation Study (outpatient group)
blood marker HbA1C (%) | 6 months
  Validation Study (outpatient group)
blood marker Fasting glucose (mmol/l) | 6 months
  Validation Study (outpatient group)
blood marker Vitamin B12 (ng/l) | 6 months
  Validation Study (outpatient group)
blood marker Folate (µg/l) | 6 months
  Validation Study (outpatient group)
blood marker Iron (µmol/l) | 6 months
  Validation Study (outpatient group)
blood marker Transferrin (µmol/l) | 6 months
  Validation Study (outpatient group)
blood marker Soluble transferrin receptor (mg/l) | 6 months
  Validation Study (outpatient group)
blood marker Ferritin (µg/l) | 6 months
  Validation Study (outpatient group)
blood marker high sensitive-CRP (mg/l) | 6 months
  Validation Study (outpatient group)
blood marker Interleukin-6 (pg/ml) | 6 months
  Validation Study (outpatient group)
Dietary patterns assessed with the eNutrition Optimizer (based on a food frequency questionnaire), MIND diet score ranging from 0 to 15 with 0=worst, 15=best ; Med Diet score ranging from 0 to 55 with 0=worst, 15=best | 6 months
  Change in diet (outpatient group)
BMI | 6 months
  Change in diet (outpatient group) and safety (outpatient group)
waist-to-hip ratio | 6 months
  Change in diet (outpatient group) and safety (outpatient group)
systolic and diastolic blood pressure | 6 months
  Change in diet (outpatient group)

CONTACTS AND LOCATIONS:
Overall Officials: Heike Bischoff-Ferrari, MD,DrPH, Principal Investigator — Center on Aging and Monbility, University of Zurich
Locations (1):
- Centre on Aging and Mobility, University of Zurich, Zurich, Canton of Zurich, Switzerland

IPD SHARING:
Plan to Share IPD: No